CLINICAL TRIAL: NCT02057224
Title: Metabolic and Cardiovascular Effects of Renal Denervation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Renal denervation has not been used as clinical method in our hospital the last two years
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Jonas Andersson, MD, PhD, Umeå University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: joan2014
Record Dates: First submitted 2014-01-29; First posted 2014-02-07 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Insulin Resistance; Hypertension
Keywords: Renal denervation; Hypertension; Insulin resistance; Adipose tissue function
MeSH Terms: conditions — Insulin Resistance; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): 15 clinical patients undergoing renal denervation
  Interventions: Procedure: Renal denervation using Medtronic Symplicity System (mono-electrode)

INTERVENTIONS:
Procedure: Renal denervation using Medtronic Symplicity System (mono-electrode) — Secondary hypertension is excluded by an extensive preoperative clinical investigation and the renal artery anatomy is visualized by computer tomography (with contrast). By cannulating the femoral artery both renal arteries are treated by a radiofrequency-catheter, 4-6 ablations in each artery.

SUMMARY:
Renal denervation has recently shown to improve glucose metabolism and insulin sensitivity in addition to reducing blood pressure. The mechanisms are however unclear. The investigators hypothesize that renal denervation alters adipose tissue function by reduced sympathetic outflow, measured by fat biopsies and markers of inflammation and insulin sensitivity. 15 clinical patients undergoing renal denervation are recruited to the study investigating anthropometry, peripheral blood samples, body composition, heart rate variability and subcutaneous fat biopsies at baseline and 6 months after renal denervation.

DETAILED DESCRIPTION:
Renal denervation, a catheter-based approach to reduce renal sympathetic afferent and efferent activity has been used successfully to treat drug-resistant hypertension. Previous studies has demonstrated a reduction of muscle sympathetic nerve activity and renal and total body noradrenaline spillover. In addition, renal denervation seems to improve glucose metabolism and insulin sensitivity, representing the first potential nonpharmaceutical approach for treating insulin resistance. However, the mechanisms are unclear. There is a clear relationship between sympathetic overactivity and insulin resistance. Activation of the sympathetic nervous systems contributes to insulin resistance and metabolic disorders and insulin itself induces sympathetic overactivity. One possible explanation to improved glucose metabolism after renal denervation is altered adipose tissue function (due to the reduction in sympathetic activity). Therefore,15 individuals undergoing renal denervation are recruited. The clinical study includes anthropometry, peripheral blood samples, body composition, heart rate variability and subcutaneous fat biopsies before renal denervation and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension
* Systolic blood pressure >160 mm Hg despite ≥3 antihypertensive drugs
* Clinical patients accepted for renal denervation

Exclusion Criteria:

* Type 1 diabetes
* Pregnancy
* Glomerular filtration rate ≤45 ml/min/1,73 m2
* Pacemaker/ICD
* Myocardial infarction/stroke the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-01; Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Adipose tissue function | 6 months after renal denervation
  Fat biopsies

SECONDARY OUTCOMES:
Heart rate variability | 6 months after renal denervation
Body composition | 6 months after renal denervation
  Measured by DXA

CONTACTS AND LOCATIONS:
Locations (1):
- Umeå University, Umeå, Sweden